CLINICAL TRIAL: NCT00756093
Title: Acute Comfort and Blurring Profile Evaluation of Marketed Lubricant Eye Drops
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: M-08-10
Record Dates: First submitted 2008-09-17; First posted 2008-09-19 (Estimated); Results first posted 2010-03-11 (Estimated); Last update posted 2012-02-02 (Estimated); Status verified 2012-01

CONDITIONS: Dry Eye
Keywords: Dry Eye, Artificial Tears,
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Polyethylene Glycols

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Systane Ultra Lubricant Eye Drops (Experimental): Systane Ultra Lubricant Eye Drops 1 drop each one time
  Interventions: Other: Systane Ultra Lubricant Eye Drops
- Optive Lubricant Eye Drops (Active Comparator): Optive Lubricant Eye Drops 1 drop each eye one time
  Interventions: Other: Optive Lubricant Eye Drops
- Blink Tears (Active Comparator): Blink Tears 1 drop each eye one time
  Interventions: Other: Blink Tears
- GenTeal Moderate Lubricant Eye Drops (Active Comparator): GenTeal Moderate Lubricant Eye Drops 1 drop each eye one time
  Interventions: Other: GenTeal Moderate Lubricant Eye Drops

INTERVENTIONS:
Other: Systane Ultra Lubricant Eye Drops — Systane Ultra Lubricant Eye Drops one drop each eye one time
  Arms: Systane Ultra Lubricant Eye Drops
Other: Optive Lubricant Eye Drops — Optive Lubricant Eye Drops one drop each eye one time
  Arms: Optive Lubricant Eye Drops
Other: Blink Tears — Blink Tears one drop each eye one time
  Arms: Blink Tears
Other: GenTeal Moderate Lubricant Eye Drops — GenTeal Moderate Lubricant Eye Drops one drop each eye one time
  Arms: GenTeal Moderate Lubricant Eye Drops

SUMMARY:
To evaluate drop comfort, acceptability and blur profile between four marketed artificial tears in dry eye patients

ELIGIBILITY:
Inclusion Criteria:

* documented diagnosis of dry eye

Exclusion Criteria:

* use of topical ocular drops within 2 hours preceding enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-09; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Alcon Call Center, Fort Worth, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 20 dry eye subjects
Pre-assignment Details: randomized, double-masked, cross-over design
Groups:
- Systane, Then Optive, Then Blink Tears, Then GenTeal Moderate: Pateints received Systane first, then Optive, then Blink Tears, then GenTeal Moderate last.
- Optive, Then Blink Tears, Then GenTeal Moderate, Then Systane: Patients received Optive first, then Blink Tears, then GenTeal Moderate, then Systane
- Blink Tears, Then GenTeal Moderate, Then Systane, Then Optive: Patients received Blink Tears first, then GenTeal Moderate, then Systane, then Optive last
- GenTeal Moderate, Then Systane, Then Optive, Then Blink Tears: Patients received GenTeal Moderate first, then Systane, then Optive, then Blink Tears last
Period: First Intervention
Arm/Group | Systane, Then Optive, Then Blink Tears, Then GenTeal Moderate | Optive, Then Blink Tears, Then GenTeal Moderate, Then Systane | Blink Tears, Then GenTeal Moderate, Then Systane, Then Optive | GenTeal Moderate, Then Systane, Then Optive, Then Blink Tears
Started | 5 | 5 | 5 | 5
Completed | 5 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0
Period: Second Intervention
Arm/Group | Systane, Then Optive, Then Blink Tears, Then GenTeal Moderate | Optive, Then Blink Tears, Then GenTeal Moderate, Then Systane | Blink Tears, Then GenTeal Moderate, Then Systane, Then Optive | GenTeal Moderate, Then Systane, Then Optive, Then Blink Tears
Started | 5 | 5 | 5 | 5
Completed | 5 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0
Period: Third Intervention
Arm/Group | Systane, Then Optive, Then Blink Tears, Then GenTeal Moderate | Optive, Then Blink Tears, Then GenTeal Moderate, Then Systane | Blink Tears, Then GenTeal Moderate, Then Systane, Then Optive | GenTeal Moderate, Then Systane, Then Optive, Then Blink Tears
Started | 5 | 5 | 5 | 5
Completed | 5 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0
Period: Fourth Intervention
Arm/Group | Systane, Then Optive, Then Blink Tears, Then GenTeal Moderate | Optive, Then Blink Tears, Then GenTeal Moderate, Then Systane | Blink Tears, Then GenTeal Moderate, Then Systane, Then Optive | GenTeal Moderate, Then Systane, Then Optive, Then Blink Tears
Started | 5 | 5 | 5 | 5
Completed | 5 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Overall Study
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 3

OUTCOME MEASURES:

1. Primary Outcome: Drop Comfort
Description: Drop comfort grading scale is a 0 to 9 scale, with 0 meaning most comfortable and 9 meaning most uncomfortable.
Time Frame: once upon instillation
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Systane Ultra Lubricant Eye Drops: Systane Ultra Lubricant Eye Drops
- Optive Lubricant Eye Drops: Optive Lubricant Eye Drops
- Blink Tears: Blink Tears
- GenTeal Moderate Lubricant Eye Drops: GenTeal Moderate Lubricant Eye Drops
Arm/Group | Systane Ultra Lubricant Eye Drops | Optive Lubricant Eye Drops | Blink Tears | GenTeal Moderate Lubricant Eye Drops
Number analyzed (Participants) | 20 | 20 | 20 | 20
units on a scale | 0.7 (1.26) | 1.05 (1.10) | 1.84 (2.19) | 1.1 (1.21)

ADVERSE EVENTS:
Arm/Group | Systane Ultra Lubricant Eye Drops | Optive Lubricant Eye Drops | Blink Tears | GenTeal Moderate Lubricant Eye Drops
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI should hold confidential, and not disclose directly or indirectly to any third party other than Contractors, the data arising out of the study. Alcon reserves the right of prior review of any publication or presentation of information related to the study.